CLINICAL TRIAL: NCT05391789
Title: Clinical Efficacy of Ulinastatin for Treatment of Sepsis With Systemic Inflammatory Response Syndrome: a Multicenter, Randomized, Double-blind, Multi Dose and Placebo-controlled Clinical Trial.
Brief Title: Clinical Efficacy of Ulinastatin for Treatment of Sepsis With Systemic Inflammatory Response Syndrome
Acronym: CURE-SepSIRS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Wen-hong Zhang, chief physician, professor, Huashan Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KY2021-924
Record Dates: First submitted 2021-12-28; First posted 2022-05-26 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis | interventions — urinastatin; Therapeutics

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- normal dose (Experimental): Patients would be given 400000 units of ulinastatin (specification: 100000 units / vial) dissolved in 50 ml of 0.9% normal saline intravenously for at least 1 hour, once every 8 hours. It is evaluated by the attending doctor every day. When the patient does not have systemic inflammatory response syndrome (SIRS), halve the dose and continue to use it for 2 days, with a total course of treatment of at least 3 days
  Interventions: Drug: Ulinastatin
- high dose (Experimental): Patients would be given 800000 units of ulinastatin (specification: 100000 units / vial) dissolved in 50 ml of 0.9% normal saline intravenously for at least 1 hour, once every 8 hours. It is evaluated by the attending doctor every day. When the patient does not have systemic inflammatory response syndrome (SIRS), halve the dose and continue to use it for 2 days, with a total course of treatment of at least 3 days
  Interventions: Drug: Ulinastatin
- placebo (Placebo Comparator): Patients would be given 50 ml of 0.9% normal saline intravenously for at least 1 hour once every 8 hours.It is evaluated by the attending doctor every day. When the patient does not have systemic inflammatory response syndrome (SIRS), continue to use it for 2 days, with a total course of treatment of at least 3 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ulinastatin — Patients would be given 400000 or 800000units of ulinastatin (specification: 100000 units / vial) dissolved in 50 ml of 0.9% normal saline intravenously for at least 1 hour, once every 8 hours. It is evaluated by the attending doctor every day. When the patient does not have systemic inflammatory response syndrome (SIRS), halve the dose and continue to use it for 2 days, with a total course of treatment of at least 3 days
  Other Names: Treatment
  Arms: high dose; normal dose
Drug: Placebo — Patients would be given 50 ml of 0.9% normal saline intravenously for at least 1 hour once every 8 hours.It is evaluated by the attending doctor every day. When the patient does not have systemic inflammatory response syndrome (SIRS), continue to use it for 2 days, with a total course of treatment of at least 3 days.
  Other Names: Control
  Arms: placebo

SUMMARY:
Sepsis is a life-threatening organ dysfunction caused by the maladjusted response of the host to infection. It is a clinical syndrome with high mortality. Studies have confirmed that many cytokines play a vital role in the pathogenesis of sepsis. Ulinastatin (UTI) is a glycoprotein that exists in human blood and can be isolated and purified from human urine. It is a broad-spectrum protease inhibitor. Previous studies have shown that Ulinastatin may have the effect of treating sepsis.

120 septic patients with systemic inflammatory response syndrome would be recruited and randomly assigned to the ordinary dose group, high dose group and placebo control group according to the ratio of 1:1:1.

The trial will be followed up on days 0, 1, 3, 5, 7 and 28. Sofa on day 7 compared with baseline and all-cause mortality on day 28 were investigated to explore the efficacy of ulinastatin in the treatment of adult sepsis patients with systemic inflammatory response syndrome.

DETAILED DESCRIPTION:
The study plans to recruit 120 septic patients with systemic inflammatory response syndrome. After signing the informed consent, they will be included as day 0. They will be randomly assigned to the ordinary dose group, high dose group and placebo control group according to the ratio of 1:1:1, and the evaluation of basic clinical information of subjects will be supplemented and improved.The ordinary dose group will receive 400000 units of ulinastatin, which will be injected intravenously every 8 hours, The high-dose group will receive 800000 units of ulinastatin intravenously every 8 hours, and the control group will use equal volume solvent (50ml normal saline) as placebo intravenously every 8 hours. When the patient does not have systemic inflammatory response syndrome, the dose will be halved and then continue to be used for 2 days. The total course of Ulinastatin injection shall be at least 3 days.

Inclusion criteria:

1) Adults ≥ 18 years old and ≤ 80 years old 2) meet the sepsis-3.0 standard specified by the American Society of critical care medicine and the European Society of critical care medicine 3) sepsis diagnosis time < 48h 4) systemic inflammatory response syndrome (SIRS) 5) obtain the informed consent signed by the patient or authorized immediate family members

Exclusion criteria:

1) Congestive heart failure, NYHA grade IV cardiac function, cerebrovascular accident or acute coronary syndrome within 3 months, cardiac arrest in this hospital or within 7 days, non infectious cardiogenic shock, uncontrolled acute bleeding 2) severe chronic liver disease (child Pugh grade C), liver parenchymal disease with significant portal hypertension Acute liver failure 3) chronic renal failure, who had received dialysis treatment before enrollment 4) severe abnormal coagulation function: isth-dic score ≥ 5 points 5) significant immune abnormalities / damage: organ or bone marrow transplantation and moderate and severe leucopenia within 3 months before screening, such as neutrophils < 1.5 × 109 / L, received radiotherapy or chemotherapy within 3 months, HIV seropositive, hematological / lymphatic system tumor active period 6) received Xuebijing, thymosin or gamma globulin treatment within 3 months before study enrollment 7) others: allergic to study drugs, pregnancy, lactation, participated in other clinical trials within 3 months, and other situations that researchers think are not suitable to participate.

The trial will be followed up on days 0, 1, 3, 5, 7 and 28. The changes of sofa on day 7 compared with baseline, all-cause mortality on day 28, ICU hospitalization time, antibiotic use time, SIRS duration, vasoactive drug time, mechanical ventilation time, CRRT time, infection and inflammation indexes, coagulation and fibrinolysis indexes, liver function, renal function, nervous and mental system function and endothelial cell function were compared, To explore the efficacy of ulinastatin in the treatment of adult sepsis patients with systemic inflammatory response syndrome.

ELIGIBILITY:
Inclusion Criteria:

1. sepsis-3 specified by SCCM and ESICM 1) suspected or confirmed infection: diagnosed by a clinician 2) evidence of acute organ dysfunction: for patients without chronic organ dysfunction in the past (assuming a baseline SOFA score of 0): sofa ≥ 2 points from 48 hours before diagnosis of infection to 24 hours after diagnosis of infection for patients with chronic organ dysfunction in the past (SOFA score should be based on baseline): the increase of sofa ≥ 2 points from 48 hours before diagnosis of infection to 24 hours after diagnosis of infection
2. diagnosis of sepsis for less than 48 hours
3. Systemic inflammatory response syndrome (SIRS) 1) body temperature > 38 ℃ or < 36 ℃ 2) heart rate > 90 3) respiratory rate> 20 4) WBC count > 12 × 10 ^ 9 / L or < 4 × 10^9/L (>12000/ μ L or < 4000/ μ L or immature granulocytes > 10%)
4. Obtained informed consent signed by the patient or authorized immediate family member

Exclusion Criteria:

1. Congestive heart failure (NYHA heart function level 4), cerebrovascular accident or acute coronary syndrome within 3 months, cardiac arrest within 7 days of this hospitalization, non-infectious cardiogenic shock, uncontrolled acute bleeding
2. Severe chronic liver disease (Child-Pugh grade C), liver parenchymal lesions with obvious portal hypertension, acute liver failure
3. Chronic renal failure, received dialysis treatment before being selected
4. Severe coagulation function: ISTH-DIC score ≥ 5 points
5. Significant immune abnormality/injury: received organ or bone marrow transplantation within 3 months before screening, moderate to severe leukopenia such as neutrophils <1.5×10^9/L, received radiotherapy or chemotherapy within 3 months , HIV seropositivity, active blood/lymphatic system tumor
6. Have received Xuebijing, thymosin or gamma globulin treatment within 3 months before being selected for the study
7. Others: allergies to study drugs, pregnancy, breast-feeding, participating in other clinical trials within 3 months, and other conditions deemed unsuitable by the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-07 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
delta sofa, ΔSOFA | Day 5
  Sequential organ failure asses(SOFA) of day 5 , compared with the baseline.

SECONDARY OUTCOMES:
Sofa vs. baseline change in sofa at randomization (delta sofa, Δ SOFA） | Day 1,3,7
  Sequential Organ Failure Assessment
28 day all-cause mortality | Day 28
  28 day all-cause mortality
ICU hospitalization days | Day 28
  ICU hospitalization days
antibiotic use days | Day 28
  antibiotic use days
SIRS days | Day 28
  SIRS days
vasoactive drugs days | Day 28
  vasoactive drugs days
mechanical ventilation days | Day 28
  mechanical ventilation days
CRRT days | Day 28
  CRRT days
Blood routine | Day 1,3,5,7
  Blood routine
coagulation and fibrinolysis indexes: PT, PLT, D-dimer | Day 1,3,5,7
  coagulation and fibrinolysis indexes
DIC score | Day 1,3,5,7
  The ISTH group produced a simple scoring system for the diagnosis of DIC depending on the Platelet count, the PT, the fibrinogen level and critically the FDP/D-Dimer results. A person's ISTH DIC score ranges from 0 to 8. <5 is suggestive of non-overt/low grade DIC. ≥5 means laboratory evidence is consistent with overt DIC
AST, ALT, bilirubin | Day 1,3,5,7
  Liver function
urine volume | Day 1,3,5,7
  urine volume
creatinine | Day 1,3,5,7
  creatinine
urea nitrogen | Day 1,3,5,7
  urea nitrogen
blood lactate | Day 1,3,5,7
  blood lactate
oxygenation index | Day 1,3,5,7
  oxygenation index
oxygen saturation | Day 1,3,5,7
  oxygen saturation
Glasgow Coma Scale | Day 1,3,5,7
  Glasgow Coma Scale. A person's GCS score can range from 3 (completely unresponsive) to 15 (responsive). A lower score means a more serious condition.
days of delirium and coma | Day 1,3,5,7
  days of delirium and coma
APACHE-II on day 5 | Day 5
  Acute Physiology and Chronic Health Evaluation
ADL on day 1,3,5,7; | Day 1,3,5,7
  Activities of Daily Living score
intercellular adhesion factor | Day 1,3,7
  Endothelial cell function
concentration of endothelial cell specific molecules | Day 1,3,7
  Endothelial cell function
heparan sulfate | Day 1,3,7
  Endothelial cell function
lymphocyte subsets and inflammatory factor levels (IL-6, IL-10, CRP, PCT, TNF- α、 HMGB-1） | Day 1,3,7
  Immune and inflammatory indexes

OTHER OUTCOMES:
adverse event | Day 28
  safety endpoint
Serious adverse events | Day 28
  safety endpoint
Vital signs | Day 28
  any abnormalities in vital signs
Blood biochemistry | Day 28
  safety endpoint
physical examination results | Day 28
  any abnormalities in physical examination results
electrocardiogram | Day 28
  any abnormalities in electrocardiogram

CONTACTS AND LOCATIONS:
Overall Officials: Wenhong Wenhong, Professor, Principal Investigator — Huashan Hospital
Locations (1):
- Huashan Hospital affiliated to Fudan University, Jingan, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No